CLINICAL TRIAL: NCT06243419
Title: The Effect Of Vein Imaging Device And Virtual Reality On Catheter Intervention Success, Procedure Related Outcomes During Peripheral Intravenous Catheterization in Children
Brief Title: Veın Imagıng Devıce And Vırtual Realıty
Acronym: ven-VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, pHD, Assoc. Prof., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ven-VR
Record Dates: First submitted 2023-05-24; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Pain, Acute; Emotional Distress; Fear; Anxiety State
MeSH Terms: conditions — Acute Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- vein viewer (Experimental): The vein imaging device was used before the vascular access attempt
  Interventions: Device: vein viewer
- virtual reality (Experimental): wearing virtual reality glasses
  Interventions: Device: virtual reality
- vein viewer and virtual reality (Experimental): The vein imaging device was used before the vascular access attempt and wearing virtual reality glasses
  Interventions: Device: vein viewer and virtual reality
- Control group (No Intervention): standard care

INTERVENTIONS:
Device: vein viewer — The PIC region was visualized with the help of the device, and the vein to which the intervention would be applied was determined.
  Arms: vein viewer
Device: virtual reality — The child watched the application by wearing virtual glasses during the PIC insertion
  Arms: virtual reality
Device: vein viewer and virtual reality — The PIC region was visualized with the help of the device, and the vein to which the intervention would be applied was determined.
  The child watched the application by wearing virtual glasses during the PIC insertion
  Arms: vein viewer and virtual reality

SUMMARY:
The aim of this study was to evaluate the effect of a vein imaging device and virtual reality distraction on the success of peripheral intravenous catheter (PIC) placement, intervention duration, emotional appearance, pain, fear, and anxiety related to PIC intervention in children aged 4-10 years in a pediatric emergency unit.

DETAILED DESCRIPTION:
The children were divided into four groups: control group, vein imaging group, virtual reality group, and vein imaging and virtual reality group. The duration of the intervention and the number of PIC interventions performed on each patient were recorded. The children were assessed before and after the procedure using the Emotional Appearance Scale for Children. After the procedure, the Child Fear Scale and Child Anxiety Scale-State were used to evaluate the most painful moment experienced by the child during the procedure using the Wong-Baker FACES (WB-FACES) and Color Analog Scale.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 4-10
* The child agrees to voluntarily participate in the study.
* Parents agree to voluntarily participate in the study
* Obtaining consent from the child and parent

Exclusion Criteria:

* Need for urgent resuscitation
* Having a fever (>37.5C) and severe dehydration
* The fact that the patient had taken analgesics before the PIC intervention.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Pain assesed by Wong-Baker FACES | immediately after the vascular access (on average 2-3 minutes later)
  Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10.
Anxiety assesed by Children Anxiety Meter-State | immediately after the vascular access (on average 2-3 minutes later)
  The Children's Anxiety Meter. The Children's Anxiety Meter assesses children's anxiety and uses before medical procedures. This scale is drawn like a thermometer with a bulb at the bottom and also includes horizontal lines at intervals going up to the top (0-10). higher scores mean a worse outcome.
Fear assesed by Child Fear Scale | immediately after the vascular access (on average 2-3 minutes later)
  The Child Fear Scale. This one-item scale measures procedure-related fear in children, consisting of five sex-neutral faces ranging from 0 (no fear) to extreme fear. This rating scale ranges from 0 to 4. It ranges from a no-fear (neutral) face (0) on the far left to a face showing extreme fear on the far right. Higher scores mean a worse outcome.
the success of peripheral intravenous catheter (PIC) placement | at PIC insertion
  first IV attempt
Emotional Appearance by Emotional Appearance Scale for Children | before the PIC insertion and immediately after the PIC insertion (on average 2-3 minutes later)]
  This scale allows direct behavioral observation, and consists of 5 different behavioral categories; 'Facial Expression', 'Speaking', 'Activity', 'Interaction' and 'Cooperation Level'. Scale scoring is done by reviewing the descriptions of behavior in each category and selecting the numerical value that most represent the observed behavior. Each category is scored from 1 to 5. The total score is made so that the numerical value is between 5-25 by adding the points obtained for each category. A higher scale score indicates the appearance of more negative emotional behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin Özalp Gerçeker, Assoc. Prof., Principal Investigator — Dokuz Eylul University
Locations (1):
- Gülçin Özalp Gerçeker, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Can M, Ozalp Gerceker G. The effect of the Veinlite PEDI2 and passive virtual reality distraction on peripheral catheter insertion-related emotional behavior, pain, fear, and anxiety of children: A randomized controlled trial. J Pediatr Nurs. 2024 Sep-Oct;78:e227-e235. doi: 10.1016/j.pedn.2024.07.010. Epub 2024 Jul 26. PMID 39060169